CLINICAL TRIAL: NCT02353195
Title: "Analgesic Effects of Capacitive Resistive Monopolar Radio-frequency (448 kHz) in Patients With Myofascial Chronic Neck Pain: A Pilot Randomized Controlled Trial."
Brief Title: Effects of Radio-frequency in Patients With Myofascial Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15/2013
Record Dates: First submitted 2015-01-27; First posted 2015-02-02 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radio-frequency group (Experimental): The equipment used, (INDIBA® activ 902, (448kHz)). The electricity was administered in the following manner: cream was applied to the site with the severe rest pain and its adjacent area, and the electrical output was increased by moving the movable electrode within the patient´s tolerance level, while monitoring the skin temperature tolerable to the patient. Therapy was conducted for 12 minutes, two times per week over four weeks (eight sessions in total)
  Interventions: Other: Radiofrequency
- Placebo group (Placebo Comparator): All patients were treated with the same device in a nonfunctional application (no energy source) and the therapy was conducted for 12 minutes, two times per week over four weeks (eight sessions in total).
  Interventions: Other: Radiofrequency

INTERVENTIONS:
Other: Radiofrequency — The equipment used, 35-mm diameter CAP and 30-mm diameter RES movable electrode was used on the affected site, and a planar electrode was used as a return electrode on the abdomen. The electricity was administered in the following manner: cream was applied to the site with the severest pain and its adjacent area, and the electrical output was increased by moving the movable electrode within the patient´s tolerance level, while monitoring the skin temperature tolerable to the patient.

SUMMARY:
The aim of this study was to evaluate the potential clinical benefits of Monopolar Capacitive Resistive Radio-frequency (448 kHz) (MCRR)F for the treatment of myofascial chronic neck pain.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled trial. Setting: University community.

Patients with myofascial chronic neck pain with active MTrP in one upper trapezius muscle were involved. The patients were randomly divided into two groups: a radiofrequency group (RFG), who (14 patients) received 8 sessions of a monopolar capacitive resistive radiofrequency (MCRRF) application over the upper trapezius muscle and ten patients received 8 sessions of placebo radiofrequency (PG) over the same muscle. Main outcome measures: Visual analog scale (VAS), neck disability index (NDI) and cervical range of motion (pre-treatment, immediately post-first session treatment and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

-Patients aged between 18 and 60 years with myofascial chronic neck pain. The area of neck pain was defined as the cervical region, possibly with referred or radiating pain into the occiput, nuchal muscles, shoulders and upper limbs. Symptoms had to have been present for at least six months before. At least one active MTrP in one upper trapezius muscle had to be present. For bilateral neck pain, the most painful side was designated for treatment.

Exclusion Criteria:

* Severe disorders of the cervical spine, such as spinal stenosis, disk prolapse, postoperative conditions of the neck and shoulder areas, history of severe trauma, whiplash, spasmodic torticollis, instability, migraine, peripheral nerve entrapment, fibromyalgia, shoulder diseases, inflammatory rheumatic diseases, severe psychiatric illness and pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS). | 1 month
  Pain intensity was measured using a 100-mm visual analogue scale (VAS). This scale consists of a 100-mm horizontal line with pain descriptors ranging from "no pain" marked on the left side to "the worst pain imaginable" on the right side. The perceived pain level of the patients was measured at rest, by marking the VAS with a perpendicular line. This is a valid method to measure pain level, and psychometric properties of the VAS have been reported widely. The minimal important difference of the VAS is based on detecting an 8.6-mm difference (based on a previous study for a score < 40 mm with a pain onset of greater than 12 weeks) immediately after treatment The VAS has been documented in previous studies as having good reliability and validity.

SECONDARY OUTCOMES:
Neck disability | 1 month
  The Neck Disability Index (NDI) was used. NDI is a self-reporting questionnaire used to determine how neck pain affects a patient's daily life. It consists of ten questions in the following domains: Pain Intensity, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, and Recreation. Each question contains six response options, scored from 0 (no disability) to 5 (complete disability). All section scores are then totaled. Scoring is reported on a 0-50 scale (0 being the best possible score and 50 the worst). The NDI has good construct validity. The NDI is seen as a valid tool to measure neck pain and disabilities in patients with neck pain due to acute or chronic conditions, as well as in patients suffering from musculoskeletal dysfunctions.
Cervical Range of Motion | 1 month
  Cervical range of movement was measured with adevice (Performance Attainment Associates, Roseville, MN) .The device was placed on the subject's head, and a magnetic collar, also part of the device, was placed on the shoulders to take into account any rotation of the trunk.a chair was used on which the subjects were sitting to kept in the same position for all data collection. The initial position of the head was set to neutral at the zero mark of the inclinometer for flexion, extensión both side flexion and rotation. Three trials were executed consecutively in each direction, and the average of the three trials was computed.

CONTACTS AND LOCATIONS:
Overall Officials: Josué Fernández-Carnero, PhD, Principal Investigator — Universidad Rey Juan Carlos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diego IMA, Fernandez-Carnero J, Val SL, Cano-de-la-Cuerda R, Calvo-Lobo C, Piedrola RM, Oliva LCL, Rueda FM. Analgesic effects of a capacitive-resistive monopolar radiofrequency in patients with myofascial chronic neck pain: a pilot randomized controlled trial. Rev Assoc Med Bras (1992). 2019 Feb;65(2):156-164. doi: 10.1590/1806-9282.65.2.156. PMID 30892438
- See also: web site of the University — http://www.urjc.es